CLINICAL TRIAL: NCT04937881
Title: Comparison of Pharmacokinetics of Tenofovir Alafenamide (TAF) With Tenofovir Disoproxil (TDF) in Pregnant and Postpartum Women and Their Infants in PrEP-PP Study
Brief Title: PK of TAF and TDF for PrEP in Pregnant and Postpartum Women
Acronym: PrEP-PP PK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Cape Town (Other); Desmond Tutu HIV Foundation (Other); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Dvora Joseph Davey, PhD, MPH, Associate Professor, Epidemiology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CO-US-412-6091
Record Dates: First submitted 2021-06-08; First posted 2021-06-24 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Hiv
Keywords: pre-exposure prophylaxis; PrEP; pregnancy; postpartum; HIV prevention; pharmacokinetics; TAF; TDF
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — tenofovir alafenamide; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: This phase III study is a randomised control trial (RCT) of up to 60 pregnant women who will be recruited at first antenatal visit (ANC) from the Gugulethu Midwife and Obstetrics Unit.
  Participants will be randomized into the TDF vs TAF arm:
  TDF Arm: Women will receive a fixed dose combination of 200 mg emtricitabine (FTC) and 300 mg tenofovir disoproxil fumarate (TDF) administered once daily under direct observation for 8 weeks during pregnancy and again for 8 weeks in postpartum period
  TAF Arm: Fixed dose combination of 200 mg emtricitabine (FTC) and 25 mg tenofovir alafenamide (TAF) administered once daily under direct observation for 8 weeks during pregnancy and again for 8 weeks in postpartum period Women will provide their own controls, providing pregnant and postpartum samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TAF arm (Experimental): Fixed dose combination of 200 mg emtricitabine (FTC) and 25 mg tenofovir alafenamide (TAF) delivered under direct observation for 8 weeks during pregnancy and 8 weeks in postpartum period
  Interventions: Drug: Tenofovir alafenamide
- TDF arm (Active Comparator): Fixed dose combination of 200 mg emtricitabine (FTC) and 300 mg tenofovir disoproxil fumarate (TDF) delivered under direct observation for 8 weeks during pregnancy and 8 weeks in postpartum period
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir alafenamide — Daily DOT fixed dose combination of 200 mg emtricitabine (FTC) and 25 mg tenofovir alafenamide (TAF)
  Other Names: TAF
  Arms: TAF arm
Drug: Tenofovir Disoproxil Fumarate — Daily DOT fixed dose combination of 200 mg emtricitabine (FTC) and 300 mg tenofovir disoproxil fumarate (TDF)
  Other Names: TDF or Truvada
  Arms: TDF arm

SUMMARY:
This study will establish benchmarks of TFV-DP concentrations as measures of adherence following daily dosing with Tenofovir Alafenamide (TAF) compared with Tenofovir Disoproxil Fumarate (TDF) during pregnancy and postpartum. Study Investigators will recruit from an ongoing observational cohort study in Cape Town, South Africa, PrEP-PP (recruitment ongoing through July, 2021; NIMH R01MH116771; PI Coates & Myer). Findings form this PK sub-study will be used to inform future PrEP in pregnancy and postpartum studies and develop benchmarks of the relative PK between TDF and TAF.

DETAILED DESCRIPTION:
This study will establish benchmarks of TFV-DP concentrations as measures of adherence following daily dosing with Tenofovir Alafenamide (TAF) compared with Tenofovir Disoproxil Fumarate (TDF) during pregnancy and postpartum. Study Investigators will recruit from an ongoing observational cohort study in Cape Town, South Africa, PrEP-PP (recruitment ongoing through July, 2021; NIMH R01MH116771; PI Coates & Myer). Findings form this PK sub-study will be used to inform future PrEP in pregnancy and postpartum studies and develop benchmarks of the relative PK between TDF and TAF.

Study aims. (1) To establish benchmarks of TFV-DP concentrations as measures of adherence following daily dosing with TAF vs TDF in pregnancy and again in postpartum; (2) To compare the difference of TFV-DP within TDF and TAF for pregnancy vs. postpartum, and to establish adherence benchmarks of levels of TFV in breastmilk in postpartum women and compare with TDF sample.

The study will take place in an urban township in Cape Town (Gugulethu) with high HIV incidence that spans the different socioeconomic, cultural, and ethnic groups in South Africa. We selected this community because of the high HIV prevalence there in pregnant and breastfeeding women, and because of the high number of mothers visiting every month for ANC and labour/delivery.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. confirmed HIV-negative (confirmed with a 4th generation antigen HIV test) at time of study entry
3. intend on giving birth in the MOU facility
4. confirmed to be 14-24 weeks pregnant
5. without psychiatric or medical contraindications to PrEP
6. estimated creatinine clearance (CrCI) >60mL/min
7. resides close to clinic (<10km)
8. has a smart phone that can take video footage (with data bundle from study)
9. agrees to provide video phone footage of taking a pill a day for 8 weeks during pregnancy and again for 8 weeks in postpartum period

Exclusion Criteria:

Individuals not meeting the above criteria or meeting any of the following criteria will be excluded:

1. Concurrent enrolment in another HIV-1 vaccine or prevention trial
2. History of renal disease
3. Current clinical diagnosis of hypertension
4. Exhibiting psychotic symptoms
5. Currently or history of taking an anti-psychotic medication
6. Positive Hepatitis B surface antigen (HBsAg) test on screening
7. History of bone fracture not related to trauma
8. Any other medical, psychiatric or social condition which in the opinion of the investigators would affect the ability to consent and/or participate in the study
9. Any maternal or fetal complication, obstetric or medical, detected during routine care or study procedures that requires referral of pregnant or postpartum women/infants to secondary or tertiary obstetric or medical care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Landon Myer, MD, Principal Investigator — UCT
Locations (1):
- Gugulethu Midwife Obstetric Unit, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2022 and October 2022, the study enrolled participants from a large, urban clinic outside of Cape Town, South Africa. Inclusion criteria required the women to: (1) be aged 18 and older; (2) test HIV-negative; (3) be between 20-30 weeks of gestation; (4) own a smart phone; and (5) to consent to daily video observations of taking a PrEP pill.
Pre-assignment Details: We received IRB approval to increase the sample size to up to 30 participants per group to account for potential attrition and pregnancy loss (total up to N=60 women).
Groups:
- TAF Arm: Fixed dose combination of 200 mg emtricitabine (FTC) and 25 mg tenofovir alafenamide (TAF) delivered under direct observation for 8 weeks during pregnancy and 8 weeks in postpartum period
  Tenofovir alafenamide: Daily DOT fixed dose combination of 200 mg emtricitabine (FTC) and 300 mg tenofovir disoproxil fumarate (TDF)
- TDF Arm: Fixed dose combination of 200 mg emtricitabine (FTC) and 300 mg tenofovir disoproxil fumarate (TDF) delivered under direct observation for 8 weeks during pregnancy and 8 weeks in postpartum period
  Tenofovir Disoproxil Fumarate: Daily DOT fixed dose combination of 200 mg emtricitabine (FTC) and 25 mg tenofovir alafenamide (TAF)
Period: Overall Study
Arm/Group | TAF Arm | TDF Arm
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: While N=60 women initially enrolled, final analysis population was N=39, as 7 individuals withdrew from study and 14 individuals were censored.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAF Arm | TDF Arm | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28 [25 to 32] | 29 [25 to 34] | 28 [25 to 34]
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: 18-25 years | 6 | 6 | 12
  Age, Categorical: >25 years | 14 | 13 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 19 | 39
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Tenofovir Diphosphate (TFV-DP) Levels in Plasma and Intracellular Levels in Pregnant Women on Daily PrEP
Description: Levels of TFV-DP (geometric mean), comparing the drugs TAF to TDF, observed in pregnancy.
  Note: Observation of daily PrEP dosing spanned 16 weeks in total, including 8 weeks during pregnancy and 8 weeks in postpartum. Once participants had completed their 8 weeks of in-pregnancy observation, observation of therapy was paused until they entered the postpartum phase.
Time Frame: 8 week period during Pregnancy
Measure: Geometric Mean (95% Confidence Interval); unit: TFV-DP PBMC (fmol/10^6cells)
Arm/Group | TAF Arm | TDF Arm
Number analyzed (Participants) | 18 | 16
TFV-DP PBMC (fmol/10^6cells) | 580 [341 to 985] | 71 [44 to 112]

2. Primary Outcome: Tenofovir Diphosphate (TFV-DP) Levels in Plasma and Intracellular Levels in Postpartum Women on Daily PrEP
Description: Levels of TFV-DP (geometric mean), comparing the drugs TAF to TDF, observed in postpartum period.
  Note: Observation of daily PrEP dosing spanned 16 weeks in total, including 8 weeks during pregnancy and 8 weeks in postpartum. Once participants had completed their 8 weeks of in-pregnancy observation, observation of therapy was paused until they entered the postpartum phase.
Time Frame: 8 week period during Postpartum (up to 1 year from baseline pregnancy visit)
Measure: Geometric Mean (95% Confidence Interval); unit: TFV-DP PBMC (fmol/10^6 cells)
Arm/Group | TAF Arm | TDF Arm
Number analyzed (Participants) | 18 | 16
TFV-DP PBMC (fmol/10^6 cells) | 666 [396 to 1123] | 73 [50 to 108]

3. Secondary Outcome: Tenofovir Diphosphate (TFV-DP) Concentrations in Plasma and Intracellular Levels Comparing Pregnancy Against Postpartum Women
Description: Plasma and intracellular concentrations of tenofovir and plasma TFV-DP in antenatal and postpartum groups intra-individual comparisons.
  Note: TFV-DP measures were obtained by DBS once a week during periods of observation. Observation of daily PrEP dosing spanned 16 weeks in total, including 8 weeks during pregnancy and 8 weeks in postpartum. Once participants had completed their 8 weeks of in-pregnancy observation, observation of therapy was paused until they entered the postpartum phase.
Time Frame: Pregnancy (TVF-DP measures via DBS collected weekly, reported 8 weeks after start of pregnancy observation); Postpartum (TVF-DP measures via DBS collected weekly, reported 8 weeks after start of postpartum observation, up to 1 year from baseline).
Measure: Median (Inter-Quartile Range); unit: TDF:fmol/3mm punch; TAF:fmol/3mm punch
Arm/Group | TAF Arm | TDF Arm
Number analyzed (Participants) | 20 | 19
TDF:fmol/3mm punch; TAF:fmol/3mm punch
  TFV-DP steady-state concentration in Pregnancy (at 8-weeks follow up via DBS) | 611.3 [396.6 to 754.5] | 410.0 [271.0 to 571.1]
  TFV-DP steady-state concentration in Postpartum (at 8-weeks follow up via DBS) | 940.5 [630.2 to 1259.3] | 518.3 [285.7 to 780.1]

ADVERSE EVENTS:
Time Frame: Participants were then observed for 16 weeks* of daily PrEP dosing *This included 8 weeks of observation during pregnancy and 8 weeks in postpartum. Once participants had completed their 8 weeks of in-pregnancy observation, observation of therapy was paused until they entered the postpartum phase. PrEP dosing was not observed or measured during this pause, but participants were supplied with sufficient pills during this time and were encouraged to continue with daily use.
Description: Serious Adverse Events, defined as any untoward occurrence that 1) results in death, 2) is life threatening, 3) requires patient hospitalization, 4) results in a congenital anomaly/ birth defect, 5) results in persistent or significant disability/incapacity, or 6) is a medically significant event or reaction, were recorded among all participants during periods of observation, according to South African Health Products Regulatory Authority (SAHPRA) safety reporting guidelines.
Arm/Group | TAF Arm | TDF Arm
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 9/20 | 5/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAF Arm (N=20) | TDF Arm (N=19)
C-Section Delivery (Emergency) (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1)
Attempted suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Intimate Partner Violence (Social circumstances) | 1 (1) | 1 (1)
Premature Birth (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Shigella dysenteriae, Infant (Infections and infestations) | 1 (1) | 0 (0)
Bartholin cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Fetal tachycardia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT04937881/Prot_SAP_000.pdf